CLINICAL TRIAL: NCT03074357
Title: Urine, DNA and Retrospective Clinical Information Collection From Patients With Alport Nephropathy.
Brief Title: Urine, DNA and Clinical Information Collection From Patients With Alport Nephropathy.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBASICHR0005
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Alport Nephropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine Saliva for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This biomarker study is a follow-up to CPLATFRM2201. The goal of CBASICHR0005 is to collect another urine sample, interval clinical information, and an optional DNA sample from as many of the original 80 patients as possible. This new information will transform the data obtained in PLATFRM2201 from a cross-section to a temporal profile, which will (a) further enable the identification of biomarkers predictive of faster progression, and (b) satisfy the FDA's recommendation to perform "natural history studies" in rare diseases.

ELIGIBILITY:
Inclusion Criteria:

• Able to communicate well with the investigator, to understand and comply with the requirements of the study and able to provide written informed consent (parent or legal guardian for pediatric and adolescent subjects), which must be obtained before any assessment is performed.

Alport Subject-Specific Inclusion Criteria:

* Participation in CPLATFRM2201
* Physically able to provide a single first-morning urine sample of at least 30 mL (one ounce). Alport patients who have initiated dialysis therapy since participation in CPLATFRM2201 are exempt from this criterion and may still participate in this study.

Healthy Volunteer-Specific Inclusion Criteria:

• Male and Female Volunteers (may include healthy siblings of Alport patients) aged 5 to 15 years.

Exclusion Criteria:

Alport Subject-Specific Exclusion Criteria:

• None

Healthy Volunteer-Specific Exclusion Criteria:

* Use of investigational drugs at the time of enrollment, or within 30 days or 5 halflives of enrollment, whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
* Known history of one of more of (a) hematuria (gross or microscopic), (b)audiological deficits, (c) fixed (non-orthostatic) proteinuria, or (d) reduced renal filtration function with serum creatinine (Cr) above the upper limit of the normal age-specific reference range, on at least 2 prior occasions (serum Cr need not be measured specifically for eligibility).
* Any other clinically significant underlying medical conditions as judged by the PI.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be males and females comprised of up to 80 Alport subjects who participated in CPLATFRM2201 study as well as up to 20 pediatric and adolescent healthy volunteers (including healthy siblings of Alport subjects) that have met all other eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Urine levels of biomarkers - corrected for urine creatinine | Day 1
  Urine levels of biomarkers, corrected for urine creatinine, in Alport subjects stratified by magnitude of proteinura.

SECONDARY OUTCOMES:
Urine level of biomarkers - corrected for urine creatinine | Day 1
  Urine levels of biomarkers, corrected for urine creatinine, in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com